CLINICAL TRIAL: NCT00417833
Title: Multifocal Electrophysiologic Findings After Intravitreal Bevacizumab(Avastin)Treatment
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor accrual
Sponsor: Asociación para Evitar la Ceguera en México (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: APEC-0017
Record Dates: First submitted 2007-01-03; First posted 2007-01-04 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Diabetic Proliferative Retinopathy; Vascular Vein Oclussion; Choroidal Neovascularization
MeSH Terms: conditions — Choroidal Neovascularization

INTERVENTIONS:
Drug: Intravitreal Bevacizumab

SUMMARY:
Purpose: Determine the short-term safety of intravitreal bevacizumab by multifocal electroretinography (mf-ERG).

Methods: 120 eyes with choroidal neovascularization, proliferative diabetic retinopathy and retinal vein occlusion received intravitreal bevacizumab (2.5mg/0.1cc). All patients underwent best corrected visual acuity, fluorescein angiography, optical coherent tomography and mf-ERG before and 1 month after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Proliferative diabetic retinopathy, vascular vein oclussion, choroidal neovascularization
* Multifocal electroretinogram before intravitreal bevacizumab and at 1,3, and 6 months after treatment
* Completely studies

Exclusion Criteria:

Complications

* Tractional Detachment
* Endophthalmitis

Sex: All
Age Groups: Child, Adult, Older Adult
Dates: Start 2005-12; Study Completion 2006-07

CONTACTS AND LOCATIONS:
Overall Officials: Myrian L Hernández, MD, Principal Investigator — Asociación para Evitar la Ceguera en México